CLINICAL TRIAL: NCT02897089
Title: Clinical Performance of Fissure Sealants Bonded With Total and Self-etch Modes of Universal Adhesive Agents
Brief Title: Effectiveness of Fissure Sealants Bonded With Different Universal Adhesives
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zafer Cavit Cehreli, DDS, PhD, Prof., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HUDHF-1
Record Dates: First submitted 2016-08-25; First posted 2016-09-13 (Estimated); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Dental Caries on Pit and Fissure Surface
Keywords: universal adhesive; fissure sealants; retention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- acid-etch (No Intervention): Acid etch+fissure sealant
- All Bond universal adhesive (Other): Acid etch+ All Bond universal adhesive agent+fissure sealant
  Interventions: Device: Adhesive agent
- All Bond universal (Other): All Bond universal adhesive agent+fissure sealant
  Interventions: Device: Adhesive agent
- Scotchbond universal adhesive (Other): Acid etch+ Scotchbond universal adhesive agent+fissure sealant
  Interventions: Device: Adhesive agent
- Scotchbond universal (Other): Scotchbond universal adhesive agent+fissure sealant
  Interventions: Device: Adhesive agent
- Clearfil universal adhesive (Other): Acid etch+ Clearfil universal adhesive agent+fissure sealant
  Interventions: Device: Adhesive agent
- Clearfil universal (Other): Clearfil universal adhesive agent+fissure sealant
  Interventions: Device: Adhesive agent
- Total-etch Dental Adhesive (Other): Acid etch+ Single Bond adhesive agent+fissure sealant
  Interventions: Device: Adhesive agent

INTERVENTIONS:
Device: Adhesive agent — Agents used to bond the restorative materials to teeth structure.
  Arms: All Bond universal; All Bond universal adhesive; Clearfil universal; Clearfil universal adhesive; Scotchbond universal; Scotchbond universal adhesive; Total-etch Dental Adhesive

SUMMARY:
The purpose of this study is to evaluate and compare the clinical retention of a resin-based fissure sealant placed with prior application of etch-and-rinse and self-etch modes of universal adhesives.

DETAILED DESCRIPTION:
Sealants will placed on previously unsealed, caries-free permanent first molars, employing a split-mouth design. 100 patients will be included the study. The teeth will be randomized into eight groups according to the adhesive systems and modes placed under the tested resin-based sealant.

Group1: Acid-Etch + Fissure sealant (ClinPro 3M ESPE, U.S.) (Control arm) Group2: All Bond Universal (Bisco Inc., Schaumburg,IL, U.S.) - with self etch technique + Fissure sealant ; Group3: All Bond Universal - total etch technique + Fissure sealant Group4: Scotchbond (Single Bond) Universal (3M ESPE, U.S.) - self etch technique + Fissure sealant Group5: Scotchbond (Single Bond) Universal - total etch technique + Fissure sealant Group6: Clearfil Universal Bond (Kuraray, Tokyo, Japan) - self etch technique + Fissure sealant Group7: Clearfil Universal Bond- total etch technique + Fissure sealant Group8: Single Bond Plus (3M ESPE)- total etch technique + Fissure sealant

Clinical assessments will be performed according to modified USPHS criteria at 3, 6, 12, 18 and 24 months. Retention, seconder caries, marginal adaptation and marginal discoloration of the sealants will be evaluated.

The data will be analyzed statistically using Fisher's Exact test and Kaplan-Meier analysis.

ELIGIBILITY:
Inclusion Criteria:

* Teeth having clinical indication of sealing with pit and fissure sealant.
* Patients with four fully-erupted permanent molars, with unstained, caries-free and unsealed pit and fissures.

Exclusion Criteria:

* Patients having incipient carious lesions, fewer erupted molars or teeth without pits on buccal/palatal surfaces.
* Patients with systemic diseases.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-03-31 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Completion of clinical evaluations (retention, secondary caries, marginal adaptation and marginal discoloration) of all teeth assessed by modified USPHS criteria | 24 months
  Long-term clinical success of different universal adhesives under fissure sealants

CONTACTS AND LOCATIONS:
Overall Officials: Zafer C Cehreli, Prof, Principal Investigator — Hacettepe University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McCafferty J, O'Connell AC. A randomised clinical trial on the use of intermediate bonding on the retention of fissure sealants in children. Int J Paediatr Dent. 2016 Mar;26(2):110-5. doi: 10.1111/ipd.12165. Epub 2015 Apr 10. PMID 25864681
- [Background] Feigal RJ, Musherure P, Gillespie B, Levy-Polack M, Quelhas I, Hebling J. Improved sealant retention with bonding agents: a clinical study of two-bottle and single-bottle systems. J Dent Res. 2000 Nov;79(11):1850-6. doi: 10.1177/00220345000790110601. PMID 11145354
- [Background] Karaman E, Yazici AR, Tuncer D, Firat E, Unluer S, Baseren M. A 48-month clinical evaluation of fissure sealants placed with different adhesive systems. Oper Dent. 2013 Jul-Aug;38(4):369-75. doi: 10.2341/12-181-C. Epub 2012 Dec 4. PMID 23210859